CLINICAL TRIAL: NCT06983366
Title: Validation and Clinical Utility of the Lung Sliding Index (LSI) for Differentiating Pulmonary Diseases: A Prospective Case-Control Study
Brief Title: Validation and Clinical Utility of the Lung Sliding Index (LSI) for Differentiating Pulmonary Diseases
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: Aliae AR Mohamed Hussein [ahussein (Unknown)
Responsible Party: Principal Investigator, Ahmad Shaddad, Associate professor of pulmonary medicine - faculty of medicine - Assuit University, Assiut University
Other Study IDs: IRBAU3211-2025
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: COPD; ILD; Bronchiectasis; Pneumothorax; Pneumonia; Pleural Effusion Disorder; Pulmonary Oedema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis; Pneumothorax; Pneumonia; Pleural Effusion; Pulmonary Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- COPD: Chronic obstructive pulmonary disease patients will be further classified as mild, moderate, severe, and very severe according to GOLD classification.
  Interventions: Diagnostic Test: Lung Ultrasound
- Pneumothorax: Patients with Pneumothorax
  Interventions: Diagnostic Test: Lung Ultrasound
- CAP: Community-acquired pneumonia will be classified using the CURB-65 score into mild, moderate, and severe.
  Interventions: Diagnostic Test: Lung Ultrasound
- ILDs: Interstitial lung diseases will be further classified using FVC% classes, categorized as mild, moderate, and severe.
  Interventions: Diagnostic Test: Lung Ultrasound
- Bronchiectasis: patients with non-cystic fibrosis bronchiectasis
  Interventions: Diagnostic Test: Lung Ultrasound
- Pleural Effusion: Patients with pleural effusion
  Interventions: Diagnostic Test: Lung Ultrasound
- Pulmonary Oedema: Patient with any degree of Pulmonary oedema
  Interventions: Diagnostic Test: Lung Ultrasound
- Control: Healthy control subjects for comparison
  Interventions: Diagnostic Test: Lung Ultrasound

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound — All enrolled patient will be subjected to Lung Ultrasound examination LUS

SUMMARY:
This upcoming case-control study aims to confirm the Lung Sliding Index (LSI), a new ultrasound score that measures how well the pleura moves, in various lung diseases. The study will check how well the LSI can tell apart different lung diseases (like pneumothorax, interstitial lung disease, COPD, pneumonia, and pulmonary edema), how it relates to signs of disease severity, and how consistent the results are between different operators who have received the same training. Secondary objectives include assessing patient and operator satisfaction and feasibility using validated Likert scales.

DETAILED DESCRIPTION:
* The study will enroll adults with various pulmonary pathologies and healthy controls. Lung ultrasound will be performed on all subjects using a standardized 12-zone protocol; each zone will be scored for pleural sliding using the LSI (0-3 per zone; total 0-36). Operator training and calibration will precede enrollment to ensure scoring consistency.
* A subset of patients will undergo repeat assessments to evaluate intra- and interobserver reliability, using independent, blinded raters.
* For correlation with LSI, we will collect clinical data, including spirometry, blood gases, symptom scores, and 6-minute walk tests. Diagnostic utility will be evaluated using ROC curves. Satisfaction and feasibility will be assessed via Likert questionnaires, with validation analyses (internal consistency, test-retest reliability).
* All data will be de-identified and securely stored. Written informed consent will be obtained from all participants.
* The study groups will include:

  1- Pneumothorax 2. Interstitial lung disease (ILD/IPF) 3. COPD/emphysema 4. Bronchiectasis 5. Community-acquired pneumonia 6. Pulmonary edema 7- Pleural effusion 8. Healthy controls
* Data Collection Methods:
* Standardized data entry forms for clinical, imaging, and outcome data.
* Centralized digital storage with access limited to study personnel.

Statistical Methods:

- Descriptive statistics for baseline data ANOVA or Kruskal-Wallis for group comparisons; post hoc testing as appropriate ROC analysis for diagnostic cut-offs Pearson/Spearman correlation for clinical associations Intraclass correlation coefficients (ICC) for reliability Cronbach's alpha for Likert scale validation Multivariable regression for confounder adjustment

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older.
* Diagnosed with one of the specified pulmonary diseases, or a healthy control
* Able to provide written informed consent

Exclusion Criteria:

* Inability to tolerate or undergo a lung ultrasound
* Extensive chest wall pathology precluding assessment
* Unscorable >2 zones per protocol
* Withdrawal of consent
* Mechanically-ventilated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years) with:
  * Pneumothorax
  * Interstitial lung disease (ILD/IPF)
  * COPD/emphysema
  * Bronchiectasis
  * Community-acquired pneumonia
  * Pulmonary edema
  * Pleural effusion
  * Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Discriminative performance of LSI (total score, 0-36) between disease groups | At Baseline
  The primary outcome is establishing a pattern of LSI among the seven studied groups

SECONDARY OUTCOMES:
Correlation of LSI with clinical severity indices | At Baseline
  Correlation of LSI with clinical severity indices (PaO₂/FiO₂ ratio, FVC %, mMRC, 6MWT)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M. Shaddad, MD, Principal Investigator — Assiut University; Aliae A. Hussien, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the decision regarding sharing individual participant data is under review and will be updated when determined